CLINICAL TRIAL: NCT05732870
Title: OSTEOMICS: Identifying Regulators of Bone Homeostasis
Acronym: OSTEOMICS
Status: Recruiting | Type: Observational
Sponsor: Relation Therapeutics (Industry)
Collaborators: Harley Street Specialist Hospital (Unknown); Fitzrovia Hospital (Unknown); Royal Free Hospital NHS Foundation Trust (Other); Bedfordshire Hospitals NHS Foundation Trust (Other); Chelsea and Westminster NHS Foundation Trust (Other); Barts & The London NHS Trust (Other); Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RRx-Profiling-001
Record Dates: First submitted 2023-01-30; First posted 2023-02-17 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Osteoporosis; Osteoarthritis; Bone Diseases; Bone Fracture; Bone Marrow Disease
MeSH Terms: conditions — Osteoporosis; Osteoarthritis; Bone Diseases; Fractures, Bone; Bone Marrow Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 10ml whole blood and discarded bone waste (generated from range of surgeries).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participant undergoing orthopaedic surgery: * Patients with osteoarthritis undergoing total joint arthroplasty, osteotomy or arthrodesis of any joint (including hip, knee, shoulder, elbow, ankle).
  * Patients with fractured neck of femurs undergoing hemiarthroplasty or total hip arthroplasty, or other internal fixation procedure.
  * Patients undergoing acute low-velocity or fragility fracture fixation surgery.
  Interventions: Procedure: Relevant orthopaedic surgery

INTERVENTIONS:
Procedure: Relevant orthopaedic surgery — Inclusion criteria is purposefully broad to examine a range of discarded bone waste. Therefore, a large number of surgical interventions are relevant.

SUMMARY:
Diseases of bone associated with ageing, including osteoporosis (OP) and osteoarthritis (OA), reduce bone mass, bone strength and joint integrity. Current non-surgical approaches are limited to pharmaceutical agents that are not disease modifying and have poor patient tolerability due to side effect profiles. Developing a fundamental understanding of cellular bone homeostasis, including how key cell types affect tissue health, and offering novel therapeutic targets for prevention of bone disease is therefore essential. This is the focus of OSTEOMICS.

A number of factors have been linked to increased risk of bone disease, including genetic predisposition, diet, smoking, ageing, autoimmune disorders and endocrine disorders. In our study, we will recruit patients undergoing elective and non-elective orthopaedic surgery and obtain surgical bone waste for analysis. This will capture a cohort of patients with bone disorders like OP and OA, in addition to patients without overt clinical bone disease. We will study the relationship between the molecular biology of bone cells, bone structure, genetics (DNA) and environmental factors with the aim of identifying and validating novel therapeutic targets.

We will leverage modern single cell technologies to understand the diversity of cell types found in bone. These technologies have now led to the characterisation of virtually every tissue in the body, however bone and bone-adjacent tissues are massively underrepresented due to the anatomical location and underlying technical challenges. Early protocols to demineralise bone and perform single cell profiling have now been developed. We will systematically scale up these efforts to observe how genetic variation at the population level leads to alterations in bone structure and quality.

Over the next 10 years, we will generate data to comprehensively characterise bone across health and disease, use machine learning to drive analysis, and experimentally validate hypotheses - which will ultimately contribute to developing the next generation of therapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with osteoarthritis undergoing total joint arthroplasty, osteotomy or arthrodesis of any joint (including hip, knee, shoulder, wrist, elbow, ankle).
2. Patient with fractured neck of femurs undergoing hemiarthroplasty or total hip arthroplasty, or other internal fixation procedure.
3. Patients undergoing acute low-velocity or fragility fracture fixation surgery.
4. Patients aged between 18-110 years old with capacity to consent.

Since deteriorating bone health including diseases like osteoporosis are primarily conditions of older age there is no practical upper age-limit. However, study involvement is limited by suitability for surgery which encompasses multiple factors considered on an individual case basis including age, frailty, comorbidities, baseline mobility, renal function and ability to consent (for instance due to dementia or delirium).

We note that our inclusion criteria is purposefully broad as we aim to deduce trends across a wide range of conditions and backgrounds.

Exclusion Criteria:

1. Patients unable to provide informed consent.
2. Patients with suspected/established underlying malignancy.
3. Patients with suspected/established osteomyelitis.
4. Patients with suspected/established bloodborne disease
5. Patients who are currently a subject of a clinical trial involving an investigational medicinal product.

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants undergoing range of orthopaedic surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Acquisition of bone waste | Within 4 hours of resection.
  Discarded bone waste to be used for the study of RNA.

SECONDARY OUTCOMES:
Acquisition of 10ml of blood. | Within 4 hours of resection.
  Discarded blood to be used for genetic sequencing, and/or other downstream omics/assays
Completion of participant questionnaire | EDC entry within 1 week of surgery.
  Patient metadata to be used to understand cohort and identify confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: Raghbir Khakha, Principal Investigator — Harley Street Specialist Hospital & Fitzrovia Hospital/QASMC; Akash Patel, Principal Investigator — Royal Free London NHS Foundation Trust; Yegappan Kalairajah, Principal Investigator — Luton & Dunstable University Hospital, Bedfordshire Hospitals NHS Foundation Trust; Victor Babu, Principal Investigator — Chelsea and Westminster NHS Foundation Trust; Jonathan Ward, Principal Investigator — Barts & The London NHS Trust; Richard Keen, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust; Ines Reichert, Principal Investigator — King's College Hospital NHS Trust
Locations (8):
- United Kingdom (8):
  - Harley Street Specialist Hospital, London, Greater London
  - Barts Health NHS Trust, London
  - Chase Farm Hospital, London
  - Fitzrovia Hospital/QASMC, London
  - King's College Hospital, London
  - Luton & Dunstable University Hospital, London
  - Royal National Orthopaedic Hospital NHS Trust, London
  - West Middlesex University Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
It is intended that the results of the study will be reported and disseminated at international conferences and in peer-reviewed scientific journals.
  When the data is no longer required by Relation Therapeutics, we may grant access to raw data (without linked identifiable patient data) and the right to publish freely. There will be no reference in the study results / reports / publications to any information that would identify participants. The final dataset, which may include a small number of select fields from the EDC database, will not contain any identifiable personal data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will not be released until the study is complete. Raw data files in the original format (e.g. fastq) and the accompanying anonymised phenotypic data will be uploaded to a public repository e.g. the NCBI database of Genotypes and Phenotypes (dbGaP) at https://www.ncbi.nlm.nih.gov/gap/.
Access Criteria: Any database selected to host genetic data must require legally-binding data access agreements with participating researchers.